CLINICAL TRIAL: NCT04694976
Title: Evaluation of Vitamin D Deficiency Distribution in Children With Sickle Cell Disease Followed in Lyon, France
Brief Title: Vitamin D Status in Children With Sickle Cell Disease Living in Lyon, France
Acronym: EVADDREP
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_0885; ID-RCB (Other: 2020-A02709-30)
Record Dates: First submitted 2020-12-31; First posted 2021-01-05 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Vitamin D Deficiency; Sickle Cell Disease
Keywords: Vitamin D deficiency prevalence rate; Vitamin D level; Children with sickle cell disease
MeSH Terms: conditions — Vitamin D Deficiency; Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sickle cell disease children from Lyon, France: Sickle cell disease children, followed in IHOPe (Institut d'Hématologie et d'Oncologie Pédiatrique) center, consulting their referring haematologist doctor or in emergency ward, with prescribed blood sample.
  Interventions: Biological: 25-OH Vitamin D measure

INTERVENTIONS:
Biological: 25-OH Vitamin D measure — As a complement to the off-study prescription, the investigator are taking two 1 mL tubes of extra blood to measure vitamin D, calcium, phosphorus, parathyroid hormone (PTH) and creatinine.

SUMMARY:
Vitamin D deficiency may be under-diagnosed in sickle cell disease French children. Therefore, the investigator need an epidemiologic study about the prevalence of vitamin D deficiency in this specific population. There are not specific guidelines neither testing nor treatment. The investigator propose to test vitamin D status in all children with sickle cell disease who are consulting their referring haematologist doctor or in the emergency ward.

ELIGIBILITY:
Inclusion Criteria:

* Children: under 18 years old
* Sickle cell any genetic type homozygous or composite heterozygous
* To receive an assessment independently of the study, during a presentation to the emergency ward and/or a follow-up consultation by the hematologist
* no parental opposition signed by at least one parent/legal representative and no child opposition
* social security beneficiary

Exclusion Criteria:

* History of hematologic grafting

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study will focus on minor patients (0-17 years) with sickle cell disease, currently monitored in the active queue of the Lyon sickle cell reference centre of IHOPe, consulting their referring physician or paediatric emergencies of HFME, and having a blood test independently of the study.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2022-02-03 (Actual); Study Completion 2022-02-03 (Actual)

PRIMARY OUTCOMES:
Determination of 25-OH Vitamin D level | Day 1
  We classify vitamin D status as follows :
  * Sufficiency > >75nmol/L (>30 ng/mL)
  * Insufficiency 50-75 nmol/L (20-30 ng/mL)
  * Deficiency 12-50nmol/L (5-20 ng/mL)
  * Severe deficiency <12 nmol/L (<5 ng/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Valérie LAUNAY, MD, Principal Investigator — Urgences pédiatriques de l'Hôpital Femme Mère Enfant - Hospices Civils de Lyon
Locations (1):
- Hôpital Femme Mère enfant - Urgences pédiatriques, Bron, France